CLINICAL TRIAL: NCT01372865
Title: A Phase III, Non-inferiority, Open-label, Multicenter and Randomized Clinical Trial About the Treatment of Mild to Moderate Persistent Allergic Rhinitis With Eurofarma Mometasone or Reference Mometasone.
Brief Title: A Clinical Trial About Treatment of Mild to Moderate Persistent Alergic Rhinnitis With Test or Reference Mometasone (PUMA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF 119
Record Dates: First submitted 2011-06-13; First posted 2011-06-14 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Mild to Moderate Persistent Allergic Rhinitis
MeSH Terms: interventions — Mometasone Furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mometasone (Experimental)
  Interventions: Drug: Mometasone furoate
- Nasonex® (Active Comparator)
  Interventions: Drug: Mometasone furoate

INTERVENTIONS:
Drug: Mometasone furoate
  Arms: Mometasone
Drug: Mometasone furoate
  Arms: Nasonex®

SUMMARY:
The primary objective will be to compare the impact of the study formulations on alergic rhinitis carriers.

ELIGIBILITY:
Inclusion Criteria:

* Sign and date the informed consent form or, in case of subjects younger than 18 years, the document must also be signed by a legal guardian;
* ≥ 12 years old;
* Suffer from mild to moderated persistent alergic rhinitis;
* Total NIS scale score ≥ 4 points at the screening visit and within at least 4 of the 7 days before the randomization visit;
* Indication for use nasal corticosteroid;
* Present with alergic rhinitis symptoms for at least 2 years;
* May undergo a washout period of at least 2 weeks

Exclusion Criteria:

* Patients with severe alergic rhinitis;
* Patients with severe co-morbidities (at the investigator's criteria);
* Patients with mild to severe persistent asthma;
* Clinical history of infection of the airways 30 days before the study entry;
* Patients with structural changes causing nasal obstruction, such as pronounced nasal septum deviation, nasal polyps or any other type of nasal malformation;
* For female subjects, be pregnant or breastfeeding or planning to become pregnant or unwilling to use safe birth control methods during the study;
* subjects in need of other drugs to treat alergic rhinitis, such as anti-immunoglobulin E, immunotherapy, anti-leukotrienes, oral corticosteroids, inhalant corticosteroids, or any administration route other than cutaneous;
* Active smokers (use of cigarette, pipe, cigar or any other form of tobacco in any amount within the past 3 months before the study entry);
* Participation in another clinical study within the past 12 months;

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Nasal Index Score (NIS) scale that evaluates nasal obstruction, coryza, and sneezing | 04 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- IMA Brasil - Instituto de Pesquisa Clínica e Medicina Avançada, São Paulo, Brazil

REFERENCES:
- [Derived] Antila MA, Castro FM, Sano F, Machado A, Fernandes F, Rosario Filho NA, Stelmach R. Mometasone furoate in the treatment of mild, moderate, or severe persistent allergic rhinitis: a non-inferiority study (PUMA). Braz J Otorhinolaryngol. 2016 Sep-Oct;82(5):580-8. doi: 10.1016/j.bjorl.2015.11.009. Epub 2016 Feb 15. PMID 26968623